CLINICAL TRIAL: NCT01989325
Title: A Study of Filanesib (ARRY-520) and Carfilzomib in Patients With Advanced Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-520-216
Record Dates: First submitted 2013-11-05; First posted 2013-11-21 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Advanced Multiple Myeloma
MeSH Terms: interventions — carfilzomib; Proteasome Inhibitors; filanesib; Dexamethasone; Steroids; Filgrastim; Granulocyte Colony-Stimulating Factor; Injections, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carfilzomib + Filanesib (Experimental): Single agent + Carfilzomib arm.
  Patients will be hydrated prior to and following carfilzomib administration and will be premedicated with dexamethasone, per the carfilzomib prescribing information.
  Filgrastim to be administered per the approved product prescribing information and institutional guidelines.
  Interventions: Drug: Carfilzomib, proteasome inhibitor; intravenous; Drug: Filanesib, KSP(Eg5) inhibitor; intravenous; Drug: Dexamethasone, steroid; oral or intravenous; Drug: Filgrastim, granulocyte-colony stimulating factor (G-CSF); subcutaneous
- Carfilzomib (Experimental): Single agent arm.
  Patients will be hydrated prior to and following carfilzomib administration and will be premedicated with dexamethasone, per the carfilzomib prescribing information.
  Interventions: Drug: Carfilzomib, proteasome inhibitor; intravenous; Drug: Dexamethasone, steroid; oral or intravenous

INTERVENTIONS:
Drug: Carfilzomib, proteasome inhibitor; intravenous — multiple dose, single schedule
Drug: Filanesib, KSP(Eg5) inhibitor; intravenous — multiple dose, single schedule
  Arms: Carfilzomib + Filanesib
Drug: Dexamethasone, steroid; oral or intravenous — as indicated, per the carfilzomib prescribing information
Drug: Filgrastim, granulocyte-colony stimulating factor (G-CSF); subcutaneous — standard of care
  Arms: Carfilzomib + Filanesib

SUMMARY:
This is a Phase 2 study during which patients with advanced multiple myeloma will receive either carfilzomib alone (single-agent) or carfilzomib in combination with investigational study drug filanesib (ARRY-520). Patients will be followed to determine the effectiveness of both single-agent carfilzomib and carfilzomib + filanesib in treating myeloma. Patients will be allowed to crossover from single-agent carfilzomib to carfilzomib + filanesib if disease progression occurs. Approximately 75 patients from the US will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed multiple myeloma with measurable disease.
* Disease refractory to last myeloma regimen.
* Patients must have received at least 2 prior treatment regimens, including bortezomib and an IMiD (e.g., lenalidomide, thalidomide, pomalidomide). Induction therapy and stem cell transplant ± maintenance are to be considered as a single regimen.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 within 14 days prior to first dose of study treatment.
* Adequate hematology, liver and renal function laboratory values within 14 days prior to first dose of study treatment.
* Additional criteria exist.

Key Exclusion Criteria:

* Prior treatment with carfilzomib, filanesib, or any other KSP inhibitor.
* Past or current plasma cell leukemia.
* Primary amyloidosis (amyloidosis associated with multiple myeloma is allowed).
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes).
* Ongoing Grade 3 or Grade 4 peripheral neuropathy, or Grade 2 peripheral neuropathy with pain despite appropriate interventions, within 28 days prior to first dose of study treatment.
* Autologous or allogeneic stem cell or bone marrow transplant within 3 months prior to first dose of study treatment.
* Concomitant malignancies or previous malignancies (other than multiple myeloma) with less than a 2-year disease-free interval at the time of first dose of study treatment. Patients with adequately resected basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or Stage 1 prostate cancer are eligible irrespective of the time of diagnosis.
* Known pulmonary hypertension of any severity.
* Concurrent cardiac disease that, in the judgment of the Investigator, would make the patient inappropriate for study participation.
* Known positive serology for the human immunodeficiency virus (HIV), active hepatitis B and/or hepatitis C.
* Acute active infection requiring treatment.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-11; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of both carfilzomib + study drug and single-agent carfilzomib in terms of progression-free survival. | 18 months

SECONDARY OUTCOMES:
Assess the efficacy of both carfilzomib + study drug and single-agent carfilzomib in terms of objective response rate. | 18 months
Assess the safety of both carfilzomib + study drug and single-agent carfilzomib in terms of adverse events, clinical laboratory tests and electrocardiograms. | 18 months
Characterize the pharmacokinetics (PK) of study drug, carfilzomib and a carfilzomib metabolite in patients treated with carfilzomib + study drug in terms of plasma concentration-time profiles and model-based PK parameters. | 6 months
Following crossover from single-agent carfilzomib, assess the efficacy of carfilzomib + study drug in terms of objective response rate. | 18 months
Following crossover from single-agent carfilzomib, assess the safety of carfilzomib + study drug in terms of adverse events, clinical laboratory tests and electrocardiograms. | 18 months

OTHER OUTCOMES:
Evaluate patient serum levels of alpha 1-acid glycoprotein (AAG) at Baseline and during the treatment period. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (22):
  - Genesis Cancer Center, Hot Springs, Arkansas
  - UCLA, Los Angeles, California
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Crescent City Research Consortium, Marrero, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Forrest General Cancer Center, Hattiesburg, Mississippi
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Memorial Sloan Kettering, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Oncology Hematology Care - Blue Ash, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Knight Cancer Institute at Oregon Health & Science University, Portland, Oregon
  - Prairie Lakes Health Care System, Watertown, South Dakota
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Simmons Cancer Center - UT Southwestern Medical Center, Dallas, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - WVU - Mary Babb Randolph Cancer Center, Morgantown, West Virginia
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests